CLINICAL TRIAL: NCT06953128
Title: Impact of General Versus Regional Anesthesia on the Incidence of Postoperative Pulmonary Complications in Peripheral Arterial Surgery: a Multicenter Randomized Clinical Trial
Brief Title: General Versus Regional Anesthesia in Peripheral Arterial Surgery
Acronym: GENERA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: Grupo Hospitalar Conceição (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 86625325.0.1001.5327
Record Dates: First submitted 2025-04-14; First posted 2025-05-01 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Postoperative Complications; Cardiovascular Diseases
Keywords: Postoperative Pulmonary Complications; Peripheral Arterial Disease; Spinal Anesthesia; General Anesthesia; Vascular Surgery
MeSH Terms: conditions — Postoperative Complications; Cardiovascular Diseases; Peripheral Arterial Disease | interventions — Anesthesia, Spinal; Anesthesia, General

STUDY DESIGN:
Intervention Model Description: Study Model Interventional (Clinical Trial) Allocation: Randomized Intervention Model: Parallel Assignment Masking: Single (Outcomes Assessor) Primary Purpose: Prevention This model reflects the trial's aim to compare two standard anesthetic strategies in parallel groups to determine which is more effective in preventing postoperative pulmonary complications after peripheral arterial revascularization.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Single-blinded (Outcomes Assessor)
  Participants and anesthesiologists will not be blinded due to the nature of the interventions (general vs. spinal anesthesia).
  However, postoperative outcome assessors and statisticians performing data analysis will be blinded to group allocation to reduce detection and assessment bias.
  Randomization will be performed using a computer-generated block sequence and managed via the REDCap platform. Allocation concealment will be maintained using sealed envelopes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Spinal Anesthesia (Experimental): Patients in this group will receive spinal (neuraxial) anesthesia with isobaric bupivacaine (15-20 mg) and intrathecal morphine (100 μg), with optional clonidine as an adjuvant. Sedation may be provided with intravenous midazolam, fentanyl, and/or propofol, as per anesthesiologist discretion. Supplemental oxygen will be administered via nasal cannula. Patients will breathe spontaneously and will not be mechanically ventilated.
  Interventions: Procedure: Spinal Anesthesia
- General Anesthesia (Active Comparator): Patients in this group will receive general anesthesia with intravenous induction (propofol or etomidate), opioids (remifentanil), and neuromuscular blockade (rocuronium), followed by endotracheal intubation and mechanical ventilation using a protective strategy (tidal volume 6-8 mL/kg predicted body weight and PEEP 5 cmH₂O). Anesthesia maintenance will include inhaled sevoflurane and continuous opioid infusion.
  Interventions: Procedure: General Anesthesia

INTERVENTIONS:
Procedure: Spinal Anesthesia — Participants will receive subarachnoid (spinal) anesthesia with 15-20 mg of isobaric bupivacaine 0.5% and 100 μg of intrathecal morphine. Clonidine (1 μg/kg) may be added at the discretion of the anesthesiologist. Sedation will be achieved with intravenous midazolam (up to 5 mg), fentanyl (up to 100 μg), and/or target-controlled infusion of propofol. Patients will remain spontaneously breathing throughout the procedure and receive supplemental oxygen via nasal cannula.
  Arms: Spinal Anesthesia
Procedure: General Anesthesia — Participants will undergo general anesthesia induced with intravenous propofol (1.5-2.5 mg/kg) or etomidate (0.2-0.3 mg/kg), remifentanil (0.2-0.4 μg/kg/min), and rocuronium (0.6 mg/kg), followed by endotracheal intubation and controlled mechanical ventilation. Maintenance will include continuous remifentanil infusion and inhaled sevoflurane. Ventilation parameters will follow a protective strategy (tidal volume 6-8 mL/kg predicted body weight and PEEP of 5 cmH₂O).
  Arms: General Anesthesia

SUMMARY:
This multicenter, prospective, randomized clinical trial aims to compare the effects of spinal (neuraxial) anesthesia with spontaneous ventilation versus general anesthesia with mechanical ventilation on the incidence of postoperative pulmonary complications in adult patients undergoing elective lower limb revascularization surgery. A total of 594 patients with symptomatic peripheral arterial disease will be randomly assigned to receive either spinal anesthesia with sedation or general anesthesia with mechanical ventilation. The primary outcome is the incidence of postoperative pulmonary complications within 30 days or until hospital discharge, including pneumonia, respiratory failure, pleural effusion, atelectasis, and other defined respiratory events. Secondary outcomes include cardiovascular events, hemodynamic instability, renal injury, delirium, extrapulmonary complications, adverse events in the operated limb, ICU and hospital length of stay, and mortality. The study will be conducted at Hospital de Clínicas de Porto Alegre, Hospital Nossa Senhora da Conceição, and other participating Brazilian centers, with an expected start date in July 2025 and completion in December 2029.

DETAILED DESCRIPTION:
This is a prospective, randomized, multicenter clinical trial designed to evaluate the impact of the anesthetic technique-general anesthesia with mechanical ventilation versus spinal (neuraxial) anesthesia with spontaneous ventilation-on the incidence of postoperative pulmonary complications in patients undergoing elective peripheral arterial revascularization surgery. The study population will include 594 adult patients (ASA II-IV) with symptomatic critical limb ischemia, scheduled for elective lower limb revascularization at tertiary hospitals in Brazil. Patients will be randomized into two groups: Group 1 will receive spinal anesthesia with intravenous sedation and supplemental nasal oxygen; Group 2 will receive general anesthesia with controlled mechanical ventilation using lung-protective strategies (tidal volume 6-8 mL/kg and PEEP 5 cmH₂O).

The primary outcome is the incidence of postoperative pulmonary complications within 30 days after surgery or until hospital discharge. These include pneumonia, respiratory failure, pleural effusion, atelectasis, pneumothorax, aspiration pneumonitis, bronchospasm, ARDS, pulmonary embolism, and exacerbation of preexisting respiratory disease, defined according to internationally recognized criteria.

Secondary outcomes include:

1. major cardiovascular complications (nonfatal myocardial infarction, acute coronary syndrome, cardiogenic shock);
2. hemodynamic complications (prolonged hypotension or distributive shock requiring vasopressors);
3. other extrapulmonary complications such as acute kidney injury, stroke, delirium, sepsis, surgical limb complications (e.g., graft thrombosis, amputation), and thromboembolic events (e.g., DVT, PE);
4. ICU and hospital length of stay, PACU time, and 30-day or in-hospital mortality.

Data collection will include perioperative gasometric evaluation, detailed intraoperative hemodynamic and ventilatory monitoring, analgesia and antiemetic usage, and adverse events tracking through predefined time points (intraoperative, immediate postoperative, and up to 30 days after surgery). Sample size calculation is based on detecting a reduction in pulmonary complications from 25% in the general anesthesia group to 15% in the spinal anesthesia group, with a power of 80% and a two-tailed alpha of 0.05. Randomization will be performed using computer-generated block sequences, and outcome assessors and statisticians will be blinded. The statistical analysis will follow the intention-to-treat principle and include regression modeling to control for potential confounders such as comorbidities and operative duration.

The study will begin in July 2025 and is expected to be completed by December 2029. Results will be published in peer-reviewed journals and used to inform perioperative management strategies in vascular surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥18 years
* ASA physical status II to IV
* Scheduled for elective peripheral arterial revascularization of the lower limbs
* Diagnosis of symptomatic peripheral arterial disease with critical limb ischemia
* Able and willing to provide informed consent

Exclusion Criteria:

* Body mass index (BMI) > 40 kg/m²
* Emergency vascular surgery
* History of lung resection surgery
* Persistent hemodynamic instability preoperatively
* History of bronchial asthma or chronic corticosteroid therapy
* History of neuromuscular disorders
* Current use of anticoagulants or antiplatelet agents contraindicating spinal anesthesia
* Contraindications to spinal anesthesia (e.g., patient refusal, infection at puncture site, increased intracranial pressure, inability to cooperate due to agitation or cognitive impairment)
* Acute vascular obstruction or other vascular complications not consistent with elective revascularization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 594 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2027-11-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Postoperative Pulmonary Complications | Up to 30 days after surgery.
  Composite incidence of pulmonary complications occurring within 30 days after surgery or until hospital discharge. Events include: pneumonia, respiratory failure, pleural effusion, atelectasis, bronchospasm, aspiration pneumonitis, pneumothorax, pulmonary embolism, exacerbation of preexisting pulmonary disease, tracheobronchitis, and acute respiratory distress syndrome (ARDS), defined according to CDC and Berlin criteria.

SECONDARY OUTCOMES:
Incidence of Major Cardiovascular Complications | Up to 30 days after surgery.
  Composite outcome including non-fatal myocardial infarction, acute coronary syndrome, and cardiogenic shock occurring in the perioperative period, defined by standard clinical and laboratory criteria.
Incidence of Hemodynamic Complications | Up to 24 hours after surgery.
  Incidence of distributive shock or persistent hypotension requiring vasopressor support during the perioperative period.
Incidence of Extrapulmonary Complications | Up to 30 days after surgery.
  Includes sepsis, acute kidney injury, delirium, stroke, venous thromboembolism, and surgical limb events (e.g., vascular graft thrombosis, ischemia, amputation), defined according to standardized criteria.
Length of Stay in Post-Anesthesia Care Unit (PACU) | Up to 30 days after surgery.
  Total number of hours from the date of surgery to hospital discharge.
30-Day Mortality | Up to 30 days after surgery.
  All-cause mortality occurring within 30 days after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Andre P Schmidt, MD, PhD, Principal Investigator — Hospital de Clínicas de Porto Alegre (HCPA)
Locations (1):
- Andre Prato Schmidt, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No
Plan to Share Individual Participant Data (IPD)? - No
  IPD Sharing Description:
  * The individual participant data (IPD) collected during the study will not be made publicly available due to ethical considerations and patient confidentiality.
  * Plan to Share IPD with Other Researchers? No
  * Available Supporting Information:
  Not applicable
  - Time Frame and Access Criteria: Not applicable

REFERENCES:
- [Background] Schmidt AP, Silvello D, Filho CTB, Bergmann D, Ferreira LEC, Nolasco MF, Pires TD, Braga WC, Andrade CF. Effects of Neuraxial or General Anesthesia on the Incidence of Postoperative Pulmonary Complications in Patients Undergoing Peripheral Vascular Surgery: A Randomized Controlled Trial. J Cardiothorac Vasc Anesth. 2025 Mar;39(3):724-732. doi: 10.1053/j.jvca.2024.12.027. Epub 2024 Dec 21. PMID 39779428
- [Background] Schmidt AP, Marques AJ, Reinstein AR, Bevilacqua Filho CT, Carmona MJC, Auler JOC Jr, Felix EA, Andrade CF. Effects of protective mechanical ventilation during general anesthesia in patients undergoing peripheral vascular surgery: A randomized controlled trial. J Clin Anesth. 2020 May;61:109656. doi: 10.1016/j.jclinane.2019.109656. Epub 2019 Nov 26. No abstract available. PMID 31784303
- [Background] Li A, Dreksler H, Nagpal SK, Brandys T, Jetty P, Dubois L, Parsons Leigh J, Stelfox HT, McIsaac DI, Roberts DJ. Outcomes After Neuraxial or Regional Anaesthesia Instead of General Anaesthesia for Lower Limb Revascularisation Surgery: A Systematic Review and Meta-Analysis of Randomised and Non-Randomised Studies. Eur J Vasc Endovasc Surg. 2023 Mar;65(3):379-390. doi: 10.1016/j.ejvs.2022.10.046. Epub 2022 Nov 3. PMID 36336286